CLINICAL TRIAL: NCT06910280
Title: Evaluation of the Feasibility of a Study Comparing Local Anesthesia and General Anesthesia in Conservative Surgery for Breast Cancer
Acronym: ESCAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2024/927
Record Dates: First submitted 2025-01-23; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; conservative surgery; local anesthesia; quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, Local; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With local anesthesia (Experimental): local anesthesia
  Interventions: Procedure: conservative surgery for breast cancer with local anesthesia
- With general anesthesia (Active Comparator): general anesthesia
  Interventions: Procedure: conservative surgery for breast cancer with general anesthesia

INTERVENTIONS:
Procedure: conservative surgery for breast cancer with local anesthesia — conservative surgery for breast cancer with local anesthesia
  Arms: With local anesthesia
Procedure: conservative surgery for breast cancer with general anesthesia — conservative surgery for breast cancer with general anesthesia
  Arms: With general anesthesia

SUMMARY:
The conservative surgery for breast cancer is the first treatment for cancer and includes :

* A partial mastectomy (removal of part of the breast)
* A sentinel lymph node analysis, depending on the case (analysis of the first lymph node(s) draining the affected breast).

This is a common procedure in the gynecology operating room, usually performed under general anesthesia. However, with surgical advancements and less invasive procedures, it has become possible and common for patients to undergo surgery in our department under local anesthesia. No data in the medical literature has yet evaluated this new anesthetic approach.

Through this study, we aim to assess the feasibility and acceptability of partial mastectomy surgery with sentinel lymph node removal under either local anesthesia or general anesthesia.

The ultimate goal of this study is to allow future patients to benefit from faster outpatient surgery, requiring less hospital stay, and to continue the progress of minimizing surgical interventions that has already been successfully undertaken in breast cancer treatment.

This is an interventional study because it involves randomization, which determines for each enrolled patient whether they will receive general anesthesia or local anesthesia. It is a feasibility and acceptability study

It is important to note that the surgery itself will not differ between the two groups: only the method of anesthesia will change. This research is being conducted at the University Hospital of Besançon and only at this center.

ELIGIBILITY:
Inclusion Criteria:

* Female over 18 years of age
* Diagnosis of invasive breast cancer (histological proof via breast biopsy)
* Tumor size less than or equal to clinical T2 according to the current cTNM classification for breast cancer"
* No clinical and/or radiological evidence of lymph node involvement
* Affiliation to a French social security scheme or beneficiary of such a scheme
* Approval in the multidisciplinary tumor board meeting for conservative treatment with partial mastectomy combined with sentinel lymph node biopsy
* Signed informed consent indicating that the patient understands the purpose and procedures required by the study and agrees to participate in the study and comply with its requirements and restrictions

Exclusion Criteria:

* Severe and morbid obesity (BMI strictly greater than 35)
* Emaciation (BMI strictly less than 18.5)
* Contraindication to the medications used in the protocol
* Contraindication to general anesthesia
* Contraindication to the local anesthesia protocol
* Tumor considered non-resectable under local anesthesia according to the surgeon's assessment
* Bifocal tumor
* Associated oncoplastic procedure
* Contralateral surgical procedure (implantable port placement, mastopexy, partial or total mastectomy)
* Withdrawal of consent prior to surgery
* Legal incapacity or limited legal capacity
* Non-fluency in the French language or poor understanding as anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* Subject currently in the exclusion period of another study or listed in the national volunteer registry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with breast cancer
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the overall feasibility of a prospective randomized two-arm protocol: 'Local Anesthesia' and 'General Anesthesia' in the context of partial mastectomy combined with sentinel lymph node study. | 2 years
  Recruitment capacity : number of women per month meeting the inclusion criteria
Evaluate the overall feasibility of a prospective randomized two-arm protocol: 'Local Anesthesia' and 'General Anesthesia' in the context of partial mastectomy combined with sentinel lymph node study. | 2 years
  Acceptability : proportion of patients who accepted inclusion in the study among those to whom it was proposed
Evaluate the overall feasibility of a prospective randomized two-arm protocol: 'Local Anesthesia' and 'General Anesthesia' in the context of partial mastectomy combined with sentinel lymph node study. | 2 years
  Adherence : proportion of women included in the study who do not withdraw their consent before the start of surgery
Evaluate the overall feasibility of a prospective randomized two-arm protocol: 'Local Anesthesia' and 'General Anesthesia' in the context of partial mastectomy combined with sentinel lymph node study. | 3 months
  Completeness : proportion of questionnaires completed at each time point of the study

SECONDARY OUTCOMES:
Describe the effectiveness and success of conservative surgery, including partial mastectomy combined with sentinel lymph node biopsy under non-tumescent local anesthesia without sedation in breast cancer | 3 months
  Proportion of surgical procedures in which the entire operative procedure could be performed under local anesthesia without the need for general anesthesia.
Quantify postoperative pain in both arms of the study | 15 days
  Numerical rating scale for pain assessment 2 hours after leaving the operating room, 24 hours after discharge from the hospital, and 15 days after the procedure. Numerical rating scale for pain assessment and DN2 score at 3 months post-procedure.
Quantify postoperative satisfaction and well-being in both arms of the study. | 3 months
  BREAST-Q - Breast Conserving Therapy Module
  Subscales of the BREAST-Q:
  Scale 6: Physical well-being: breast (preoperative) Scale 7: Physical well-being: breast (postoperative)
Describe the oncological, anesthetic, and surgical safety of the surgical procedure in both arms of the study. | 3 months
  Need for reoperation of the breast (margins considered positive in case of 'at ink' involvement [tumor in contact with the ink] for the infiltrative component and possibly associated in situ component) Need for reoperation of the axillary region Allergic reactions Other side effects related to general or local anesthesia Postoperative surgical complications (hematoma, abscess, wound dehiscence) Length of hospital stay Death

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besancon, Besançon, Franche Comte, France

REFERENCES:
- [Background] Seror J, Hequet D, Gout-Duracher C, Cittanova M laure. Faisabilité et impact de la chirurgie mammaire conservatrice sous anesthésie locale. Communication orale, Congrè SFSPM; 2022.
- [Background] Karanlik H, Kilic B, Yildirim I, Bademler S, Ozgur I, Ilhan B, Onder S. Breast-Conserving Surgery Under Local Anesthesia in Elderly Patients with Severe Cardiorespiratory Comorbidities: A Hospital-Based Case-Control Study. Breast Care (Basel). 2017 Mar;12(1):29-33. doi: 10.1159/000455003. Epub 2017 Feb 8. PMID 28611538
- [Background] Hirokawa T, Kinoshita T, Nagao T, Hojo T. A clinical trial of curative surgery under local anesthesia for early breast cancer. Breast J. 2012 Mar-Apr;18(2):195-7. doi: 10.1111/j.1524-4741.2011.01221.x. Epub 2012 Feb 2. No abstract available. PMID 22300192
- [Background] Carlson GW. Total mastectomy under local anesthesia: the tumescent technique. Breast J. 2005 Mar-Apr;11(2):100-2. doi: 10.1111/j.1075-122X.2005.21536.x. PMID 15730454
- [Background] Sleth JC, Lavie M, Mion P, Saizy C, Servais R. [Tumescent local anaesthesia for mastectomy: lidocaine plasma concentration]. Ann Fr Anesth Reanim. 2006 Jan;25(1):74-6. doi: 10.1016/j.annfar.2005.07.074. Epub 2005 Oct 26. No abstract available. French. PMID 16256296
- [Background] Saint-Roch P. L'anesthésie locale tumescente a-t-elle une place ? 2013;
- [Background] Anne-Pauline Cungi. Étude Hypno-Séno : anesthésie générale versus hypno-tumescence en chirurgie mammaire conservatrice : évaluation de la qualité des marges de résection chirurgicale. 2020;
- [Background] Sleth JC, Servais R, Saizy C. [Tumescent infiltrative anaesthesia for mastectomy: about six cases]. Ann Fr Anesth Reanim. 2008 Nov;27(11):941-4. doi: 10.1016/j.annfar.2008.08.011. Epub 2008 Nov 11. French. PMID 19004607
- [Background] Ceccarino R, Di Micco R, Cappelletti R. Aesthetic Breast Surgery Under Cold Tumescent Anesthesia: Feasibility and Safety in Outpatient Clinic. Ann Plast Surg. 2019 Oct;83(4):384-387. doi: 10.1097/SAP.0000000000001798. PMID 31524728
- [Background] Boeer B, Helms G, Pasternak J, Roehm C, Kofler L, Haefner HM, Moehrle M, Heim E, Fischer H, Brucker SY, Hahn M. Back to the future: breast surgery with tumescent local anesthesia (TLA)? Arch Gynecol Obstet. 2023 Sep;308(3):935-940. doi: 10.1007/s00404-023-06938-5. Epub 2023 Mar 6. PMID 36872392
- [Background] Groetelaers RP, van Berlo CL, Nijhuis PH, Schapers RF, Gerritsen HA. Axillary recurrences after negative sentinel lymph node biopsy under local anaesthesia for breast cancer: a follow-up study after 5 years. Eur J Surg Oncol. 2009 Feb;35(2):159-63. doi: 10.1016/j.ejso.2008.07.017. Epub 2008 Sep 11. PMID 18789841
- [Background] van Berlo CL, Hess DA, Nijhuis PA, Leys E, Gerritsen HA, Schapers RF. Ambulatory sentinel node biopsy under local anaesthesia for patients with early breast cancer. Eur J Surg Oncol. 2003 May;29(4):383-5. doi: 10.1053/ejso.2002.1420. PMID 12711294
- [Background] Luini A, Gatti G, Frasson A, Naninato P, Magalotti C, Arnone P, Viale G, Pruneri G, Galimberti V, De Cicco C, Veronesi U. Sentinel lymph node biopsy performed with local anesthesia in patients with early-stage breast carcinoma. Arch Surg. 2002 Oct;137(10):1157-60. doi: 10.1001/archsurg.137.10.1157. PMID 12361425
- [Background] Luini A, Caldarella P, Gatti G, Veronesi P, Vento AR, Naninato P, Arnone P, Sangalli C, Brenelli F, Sosnovskikh I, Peradze N, Dussan Luberth CA, Viale G, Paganelli G. The sentinel node biopsy under local anesthesia in breast cancer: advantages and problems, how the technique influenced the activity of a breast surgery department; update from the European Institute of Oncology with more than 1000 cases. Breast. 2007 Oct;16(5):527-32. doi: 10.1016/j.breast.2007.04.003. PMID 17916496
- [Background] Luini A, Gatti G, Zurrida S, Galimberti V, Paganelli G, Naninato P, Caldarella P, Rotmensz N, Winnikow E, Viale G. The sentinel lymph node biopsy under local anesthesia in breast carcinoma: experience of the European Institute of Oncology and impact on quality of life. Breast Cancer Res Treat. 2005 Jan;89(1):69-74. doi: 10.1007/s10549-004-1473-y. PMID 15666199
- [Background] Kongdan Y, Chirappapha P, Lertsithichai P. Effectiveness and reliability of sentinel lymph node biopsy under local anesthesia for breast cancer. Breast. 2008 Oct;17(5):528-31. doi: 10.1016/j.breast.2008.04.003. Epub 2008 Jun 2. PMID 18515105
- [Background] Gauthier T, Garuchet-Bigot A, Mollard J, Aubard Y. [How I... remove axillary sentinel lymph node under local anesthesia]. Gynecol Obstet Fertil. 2010 Jun;38(6):418-9. doi: 10.1016/j.gyobfe.2010.04.004. Epub 2010 Jun 4. No abstract available. French. PMID 20576555
- [Background] Fenaroli P, Tondini C, Motta T, Virotta G, Personeni A. Axillary sentinel node biopsy under local anaesthesia in early breast cancer. Ann Oncol. 2000 Dec;11(12):1617-8. doi: 10.1093/oxfordjournals.annonc.a010407. No abstract available. PMID 11205475
- [Background] Institut national du cancer. Traitements locorégionaux des cancers du sein infiltrants non métastatiques / Synthèse, collection Recomman- dations et référentiels. 2022.
- [Background] HAS. Haute Autorité de Santé. Infracyanine (vert d'indocyanine monopic) - Repérage peropératoire du ganglion sentinelle. 2022.
- [Background] Lucas N, Interne SB, Laine P, Nicolie B, Fondrinier E. [Anaphylactic shock due to patent blue: four case report and review of literature]. J Gynecol Obstet Biol Reprod (Paris). 2010 Apr;39(2):116-20. doi: 10.1016/j.jgyn.2009.10.006. Epub 2010 Jan 15. French. PMID 20079974
- [Background] C. Ngô, C. Nos, A.-S. Bats, C. Bensaid, F. Lécuru. Chirurgie locorégional des cancers du sein. In: Encyclopédie Médico-chirurgicale. Elsevier-Masson. 2020.
- [Background] Modi S, Saura C, Yamashita T, Park YH, Kim SB, Tamura K, Andre F, Iwata H, Ito Y, Tsurutani J, Sohn J, Denduluri N, Perrin C, Aogi K, Tokunaga E, Im SA, Lee KS, Hurvitz SA, Cortes J, Lee C, Chen S, Zhang L, Shahidi J, Yver A, Krop I; DESTINY-Breast01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):610-621. doi: 10.1056/NEJMoa1914510. Epub 2019 Dec 11. PMID 31825192